CLINICAL TRIAL: NCT02452645
Title: Improving Nutrition and Physical Activity Environments in Home-based Child Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brown University (Other)
Collaborators: University of Connecticut (Other); University of Rhode Island (Other); University of North Carolina (Other)
Responsible Party: Principal Investigator, Patricia M. Risica, Assistant Professor (Research) of Epidemiology, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BrownMC
Record Dates: First submitted 2015-03-30; First posted 2015-05-22 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Family Child Care Homes
Keywords: Food; Nutrition; Physical Activity; Family; Child Care; Home; Environment
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): The intervention will integrate: a) support from peer counselors with child care experience who will serve as team leaders for groups of FCCPs; b) tailored print and video materials; and c) a set of portable active toys to elicit changes to the nutrition and physical activity environments of family child care homes.
  Interventions: Behavioral: Healthy Food and Physical Activity Environments
- Comparison (Active Comparator): The comparison intervention will provide print materials and videos on literacy and school readiness to children and books in both English and Spanish. Participants will also receive support from peer counselors with child care experience.
  Interventions: Behavioral: Comparison Group

INTERVENTIONS:
Behavioral: Healthy Food and Physical Activity Environments — Tailored written materials, videos, telephone counseling, active toys
  Arms: Intervention
Behavioral: Comparison Group — Written materials, videos, books, and telephone counseling.
  Arms: Comparison

SUMMARY:
Drs. Patricia Risica (Brown University) and Kim Gans (University of Connecticut) are Dual Principal Investigators for this project. The research team will first conduct formative research using focus groups and key-informant interviews of Family Child Care Home (FCCH) providers. This formative work will inform our adaptation of components of previous evidence-based interventions to create a new innovative intervention in both English and Spanish to improve food and PA environments of Family Child Care Homes (FCCH). The intervention will integrate: a) support from peer counselors with child care experience who will serve as team leaders for groups of FCCPs; b) tailored print and video materials; and c) a set of portable active toys. A cluster-randomized trial with 132 FCCH will evaluate the effectiveness of the intervention with a Steering Committee and Community Advisory Board guiding all aspects. The Specific Aims of the study are to: 1) Conduct formative research to inform the development and adaptation of the FCCH intervention. 2) Conduct a cluster-randomized trial of the intervention's efficacy with 66 FCCH providers and a control intervention with 66 demographically-matched FCCH providers to evaluate its impact on: a) Children's overall dietary quality at FCCHs; b) Children's PA and sedentary behaviors at FCCHs; and c) the physical and social food and PA environments of FCCHs. Evaluation methods will include survey data collection of the FCCH Providers; observation of children's' dietary intake and physical activity in FCCHs; recruitment of children within the FCCH for physical and survey measurement with permission from their parents.

DETAILED DESCRIPTION:
Preschool years are critical times when dietary and PA behaviors are established and over 70% of U. S. children under the age of six attend out-of-home child care. Unhealthy food and PA behaviors contribute to the high prevalence rates of childhood obesity. Through this research study, our team will first conduct formative research using focus groups and key-informant interviews of Family Child Care Home (FCCH) providers. Partnering with Ready to Learn Providence the investigators will recruit FCCH providers to participate. The investigators will partner with Alison Tovar, PhD, (URI faculty) and her students to conduct interviews and discussion groups in English and Spanish. This formative work will inform our adaptation of components of previous evidence-based interventions to create a new innovative intervention in both English and Spanish to improve food and PA environments of Family Child Care Homes (FCCH). The intervention will integrate: a) support from peer counselors with child care experience who will serve as team leaders for groups of FCCPs; b) tailored print and video materials; and c) a set of portable active toys. A cluster-randomized trial with 132 FCCH and 396 children in their care will evaluate the effectiveness of the intervention with a Steering Committee and Community Advisory Board guiding all aspects.

The Specific Aims of the study are to: 1) Conduct formative research to inform the development and adaptation of the FCCH intervention. 2) Conduct a cluster-randomized trial of the intervention's efficacy with 66 FCCH providers and a control intervention with 66 demographically-matched FCCH providers to evaluate its impact on: a) Children's overall dietary quality at FCCHs; b) Children's PA and sedentary behaviors at FCCHs; and c) the physical and social food and PA environments of FCCHs. Evaluation methods will include survey data collection of the FCCH Providers; observation of children's' dietary intake and physical activity in FCCHs(Partnering with Diane Ward, PhD (UNC faculty) and her student/staff member team); recruitment of children within the FCCH for physical and survey measurement with permission from their parents.

The investigators will also conduct extensive mixed-methods process evaluation to determine fidelity, dose, acceptability, context, and unintended consequences; explore the relationship between outcome measures and intervention dose as well as with mediating/moderating variables, and explore the intervention effect on child BMI. If proven effective, this intervention has the potential to be replicated and widely disseminated throughout RI and the US, where improvements in the childcare environment are a high priority.

ELIGIBILITY:
Inclusion Criteria:

* operator of a FCCH
* have at least 1 children in their care,
* provide at least 2 meals/snacks to the children
* ability to read and speak English or Spanish
* expect to be in operation in a year
* have a working phone
* have either a DVD player or internet access through computer or phone

Exclusion Criteria:

* under 18 years of age
* has no children in their care between the ages of 2 and 5 years old
* child care will be closed for more than 1 month at a time in the forthcoming year.
* does not prepare the food served by the children (children bring it from home).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Change in Observed Child Dietary Intake | 8 Months
  Child food intake will be observed and recorded by trained research assistants on two days; data will be used to calculate mean daily intake of several nutrients for each child.
Change in Measured Child Physical Activity in Child Care | 8 months
  Physical activity will be measured on two days using accelerometer devices attached onto waist bands; data will be used to calculate mean energy expenditure for each child.
Change in Observed Child Dietary Intake | 12 Months
  Child food intake will be observed and recorded by trained research assistants on two days; data will be used to calculate mean daily intake of several nutrients for each child.
Change in Measured Child Physical Activity in Child Care | 12 Months
  Child food intake will be observed and recorded by trained research assistants on two days; data will be used to calculate mean daily intake of several nutrients for each child.

SECONDARY OUTCOMES:
Change in Self Reported Provider Changes in motivators | 8 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in motivators | 12 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in self-efficacy | 8 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in self-efficacy | 12 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in barriers | 8 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in barriers | 12 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in social support | 8 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in social support | 12 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in attitudes | 8 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in attitudes | 12 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in practices | 8 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in practices | 12 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in beliefs | 8 months
  These data will be collected via telephone survey of the providers.
Change in Self Reported Provider Changes in beliefs | 12 months
  These data will be collected via telephone survey of the providers.
Change in measured food and physical activity environment of the family child care home as measured by the EPAO. | 8 months
  The EPAO estimates the food and activity environment using a questionnaire completed by the trained RA regarding observed environments and practices in the family child care home throughout one day.
Measured food and physical activity environment of the family child care home as measured by the EPAO. | 12 months
  The EPAO estimates the food and activity environment using a questionnaire completed by the trained RA regarding observed environments and practices in the family child care home throughout one day.

CONTACTS AND LOCATIONS:
Locations (1):
- Ready 2 Learn, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Gans KM, Tovar A, Kang A, Ward DS, Stowers KC, von Ash T, Dionne L, Papandonatos GD, Mena N, Jiang Q, Risica PM. A multi-component tailored intervention in family childcare homes improves diet quality and sedentary behavior of preschool children compared to an attention control: results from the Healthy Start-Comienzos Sanos cluster randomized trial. Int J Behav Nutr Phys Act. 2022 Apr 15;19(1):45. doi: 10.1186/s12966-022-01272-6. PMID 35428298
- [Derived] Gans KM, Jiang Q, Tovar A, Kang A, McCardle M, Risica PM. Physical Activity and Screen Time Practices of Family Child Care Providers: Do They Meet Best Practice Guidelines? Child Obes. 2022 Jun;18(4):281-290. doi: 10.1089/chi.2021.0094. Epub 2021 Dec 1. PMID 34851731
- [Derived] Risica PM, Tovar A, Palomo V, Dionne L, Mena N, Magid K, Ward DS, Gans KM. Improving nutrition and physical activity environments of family child care homes: the rationale, design and study protocol of the 'Healthy Start/Comienzos Sanos' cluster randomized trial. BMC Public Health. 2019 Apr 18;19(1):419. doi: 10.1186/s12889-019-6704-6. PMID 30999881
- [Derived] Gans KM, Tovar A, Jiang Q, Mello J, Dionne L, Kang A, Mena NZ, Palomo V, Risica PM. Nutrition-Related Practices of Family Child Care Providers and Differences by Ethnicity. Child Obes. 2019 Apr;15(3):167-184. doi: 10.1089/chi.2018.0083. Epub 2019 Feb 1. PMID 30707598